CLINICAL TRIAL: NCT07003607
Title: Wearable Device and Self-Regulation Strategies to Promote Physical Activity Among Children With Cancer: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ke Liu (Other)
Collaborators: Sun Yat-sen University Cancer Centre (Unknown)
Responsible Party: Sponsor-Investigator, Ke Liu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: L2023SYSU-HL-025; 2024-FXY-299-Peds Onc (Other: Sun Yat-Sen University Cancer Center)
Record Dates: First submitted 2025-05-17; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: physical activity; childhood cancer; quality of life; physical activity self-efficacy; Integrated theory of health behavior change
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Smart wristband to track daily steps, followed a personalized exercise plan, and received weekly guidance
  Interventions: Behavioral: In-Hospital Program; Behavioral: Post-Discharge Program
- Control group (Placebo Comparator): Routine health education
  Interventions: Behavioral: Control group (placebo)

INTERVENTIONS:
Behavioral: Control group (placebo) — Children in the control group received routine health education, which included cancer-related treatment, care, and general health education (e.g., treatment-related, diet, and exercise) without systematic PA health education. Every four weeks, knowledge related to sports activities, the harms of insufficient physical activity, and the benefits of increasing physical activity were pushed through the WeChat platform. During the hospitalization of the child patient, they can voluntarily participate in the activities organized by social workers.
  Arms: Control group
Behavioral: In-Hospital Program — Researchers will conduct a comprehensive evaluation for each pediatric patient, including:
  * Disease status and clinical characteristics
  * Patient and family knowledge regarding physical activity (PA)
  * Availability of social support systems
  Arms: Experimental group
Behavioral: In-Hospital Program — Based on assessment findings, two structured educational sessions (20-30 minutes each) will be delivered, covering:
  * Disease-specific knowledge and PA guidelines
  * Practical strategies for safe exercise (e.g., intensity adjustment, injury prevention)
  * Interactive demonstrations of age-appropriate movement techniques
  Arms: Experimental group
Behavioral: In-Hospital Program — Patients will co-develop personalized PA plans using the six-step self-regulation framework from the ITHBC (Integrative Theory of Health Behavior Change), including:
  * Short/long-term goal formulation
  * Progress monitoring tools
  * Barrier problem-solving protocols
  Arms: Experimental group
Behavioral: Post-Discharge Program — Patients will perform PA 3-5 times weekly (20-30 minutes/session) aligned with individualized goals, adhering to oncology-specific safety guidelines
  Arms: Experimental group
Behavioral: Post-Discharge Program — Mondays: Curated PA educational content (e.g., home-based exercise videos, fatigue management tips) will be disseminated via the WeChat platform.
  Sundays: Scheduled telehealth check-ins with patients and caregivers to:
  * Review PA adherence and experiential feedback
  * Address knowledge gaps through tailored coaching
  * Reinforce behavior change techniques (e.g., self-monitoring logs)
  Arms: Experimental group
Behavioral: Post-Discharge Program — Regular monitoring and evaluation will be conducted to assess PA outcomes: comprehensive evaluations will identify barriers (e.g., treatment-related fatigue) and guide real-time adjustments to the exercise plan based on the patient's physical condition and performance. To enhance adherence, families will collaboratively set alarm reminders for PA sessions, and caregivers will be invited to supervise daily activities.
  Arms: Experimental group

SUMMARY:
This is a clinical trial that tested whether a 12-week exercise program using smart wristbands and personalized goal-setting could help children with cancer become more active, feel more confident about exercising, and improve their quality of life.

The study included 72 children and teenagers (ages 6-18) receiving cancer treatment at two hospitals in China. They were divided into two groups:

Intervention group (33 children): Used a smart wristband to track daily steps, followed a personalized exercise plan, and received weekly guidance.

Control group (39 children): Continued with usual care (no special exercise program).

The main questions it aims to answer are:

1. Does the exercise program help children with cancer move more and sit less;
2. Can it boost their confidence to stay active and improve their physical and emotional well-being?

DETAILED DESCRIPTION:
What did the study find?

* Children in the exercise group:

  * Increased active time: They did more moderate-to-vigorous exercise (like brisk walking or playing) by the end of the program.
  * Walked more steps daily: From about 2,200 steps/day at the start to over 6,300 steps/day after 12 weeks.
  * Felt more confident: They believed they could keep exercising even during treatment.
  * Improved well-being: Parents and children reported better physical energy, mood, and social interactions.
* Comparison with the control group:

  * The exercise group showed much greater improvements than the group without the program.

What does this mean for families? This study suggests that combining wearable devices (like step trackers) with simple goal-setting and family support may help children with cancer stay active during treatment. Staying active could reduce fatigue, improve mood, and support recovery.

What's next? While these results are promising, larger studies are needed to confirm the long-term benefits and safety of such programs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 18 years old;
* Children diagnosed with leukemia, lymphoma, or solid tumor confirmed by pathology or bone marrow examination;
* Obtaining informed consent from the child and their guardian;
* Approval from the attending physician for participation in physical activity interventions.

Exclusion Criteria:

* Children diagnosed with mental health disorders;
* Individuals with severe physical disabilities incompatible with physical activity participation;
* Cases involving metastasis to bone tissue that would restrict movement.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
physical activity | From enrollment to the end of treatment at 12 weeks
  This study assessed physical activity (PA) patterns in children with cancer using the Children's Leisure Time Activities Study Survey-Chinese version (CLASS-C), a culturally adapted instrument developed by thVigorous PA (e.g., running, basketballe Chinese University of Hong Kong through rigorous forward-backward translation and validation. The CLASS-C captures time spent in specific activities over the past 7 days through 21 items, recording frequency (e.g., days/week) and duration (minutes/session) across three intensity categories：Light PA (e.g., walking, stretching); Moderate PA (e.g., cycling, dancing).

SECONDARY OUTCOMES:
physical activity self-efficacy | From enrollment to the end of treatment at 12 weeks
  Physical activity (PA) self-efficacy in children with cancer was evaluated using the Chinese Short Version of the Physical Activity Self-Efficacy Scale (SPASES-C), a culturally adapted instrument derived from the original 8-item SPASES through rigorous forward-backward translation and psychometric validation. The SPASES-C assesses confidence in overcoming barriers to PA via 7 Likert-type items scored from 1 ("not confident at all") to 4 ("very confident"), yielding a total range of 7-28 points. Higher total scores reflect stronger self-efficacy beliefs (e.g., 7 = minimal confidence, 28 = maximal confidence). Internal consistency (Cronbach's α = 0.87) and construct validity (CFI = 0.93) were established in pediatric populations through prior studies.
quality of life of children with cancer | From enrollment to the end of treatment at 12 weeks
  This study utilized the Pediatric Quality of Life Inventory™ Generic Core Scales Version 4.0 (PedsQL™ 4.0 Generic Core Scales) to assess the quality of life (QoL) in children diagnosed with cancer. The PedsQL™ 4.0 is a widely validated instrument designed to measure core dimensions of health-related quality of life in pediatric populations aged 2 to 18 years, including physical, emotional, social, and school functioning. Each item is scored on a 5-point Likert scale (0 = never a problem; 4 = almost always a problem), which is then reverse-scored and linearly transformed to a 0-100 scale, where higher scores indicate better quality of life. Thus, the total score as well as subscale scores range from 0 (worst QoL) to 100 (best QoL), with higher values reflecting fewer problems and greater perceived well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Prevention Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared due to ethical restrictions protecting participant privacy, institutional data governance policies, and the absence of explicit consent for public data sharing in the original study protocol

REFERENCES:
- [Background] Atun R, Bhakta N, Denburg A, Frazier AL, Friedrich P, Gupta S, Lam CG, Ward ZJ, Yeh JM, Allemani C, Coleman MP, Di Carlo V, Loucaides E, Fitchett E, Girardi F, Horton SE, Bray F, Steliarova-Foucher E, Sullivan R, Aitken JF, Banavali S, Binagwaho A, Alcasabas P, Antillon F, Arora RS, Barr RD, Bouffet E, Challinor J, Fuentes-Alabi S, Gross T, Hagander L, Hoffman RI, Herrera C, Kutluk T, Marcus KJ, Moreira C, Pritchard-Jones K, Ramirez O, Renner L, Robison LL, Shalkow J, Sung L, Yeoh A, Rodriguez-Galindo C. Sustainable care for children with cancer: a Lancet Oncology Commission. Lancet Oncol. 2020 Apr;21(4):e185-e224. doi: 10.1016/S1470-2045(20)30022-X. PMID 32240612
- [Result] Hudson MM, Ness KK, Gurney JG, Mulrooney DA, Chemaitilly W, Krull KR, Green DM, Armstrong GT, Nottage KA, Jones KE, Sklar CA, Srivastava DK, Robison LL. Clinical ascertainment of health outcomes among adults treated for childhood cancer. JAMA. 2013 Jun 12;309(22):2371-2381. doi: 10.1001/jama.2013.6296. PMID 23757085